CLINICAL TRIAL: NCT04130256
Title: Electronic Pill Bottle Monitoring to Promote Medication Adherence for People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Multiple Sclerosis Society (Other); Pillsy, Inc. (Unknown)
Responsible Party: Principal Investigator, Farrah Mateen, Associate Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018P001820
Record Dates: First submitted 2019-10-16; First posted 2019-10-17 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
Keywords: Medication adherence
MeSH Terms: conditions — Multiple Sclerosis; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Reminders (Experimental): 43 patients, each assigned to use the electronic pill bottle for 90 days. Participants will use the bottle to house their multiple sclerosis medication. The electronic pill bottle will provide daily medication reminders for participants to take their pill.
  Interventions: Device: Electronic Pill Bottle
- Passive Adherence Monitoring (Experimental): 42 patients, each assigned to use the electronic pill bottle for 90 days. Participants will use the bottle to house their multiple sclerosis medication. The electronic pill bottle will not provide medication reminders and will only track medication use.
  Interventions: Device: Electronic Pill Bottle

INTERVENTIONS:
Device: Electronic Pill Bottle — Electronic bottles that can beep and blink to send medication use reminders, record medication use data, and upload medication use data to a secure server.
  Other Names: Pillsy

SUMMARY:
People with multiple sclerosis (MS) have variable adherence to MS medications, making the full efficacy of disease modifying therapies unrealized and the assessment of true treatment failures challenging. Whereas some patients forget to take medications due to active lifestyles, others may have cognitive impairments that prevent them from organizing and planning their regular dosing schedules. An electronic pill cap ("Pillsy") has been developed to record pill taking, timing, and set reminders through a mobile app. Data on adherence can be captured and analyzed remotely for health care provider review.

DETAILED DESCRIPTION:
The investigators will enroll 85 adult patients, 18 years old and above, with relapsing remitting multiple sclerosis (RRMS), at the Massachusetts General Hospital MS Clinics in a pilot study of Pillsy electronic pill bottles. People with RRMS who are taking (1) fingolimod, (2) dimethyl fumarate, (3) terifluonomide, (4) diroximel fumarate, or (5) siponimod will be eligible. Patients must possess any type of smartphone capable of downloading the Pillsy application to be eligible. Per the Pillsy manufacturer, the Pillsy application is available on iPhones connected to the Apple App Store and smartphones running the Android operating system that are connected to the Google Play Store. Participants will be asked to use the Pillsy bottle for 90 days each. Participants will be randomized 1:1 to two conditions: 1) active reminders and 2) passive adherence tracking. Patients in the active reminders group will receive daily alerts through the Pillsy bottle, the Pillsy app, and their phone to remind them to take their pill. Patients in the passive adherence tracking group will not receive reminders and will instead have usual adherence monitored by the electronic pill bottle.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide individual written consent
* Ability to understand sufficient levels of English to use the Pillsy app
* Ability to come to Massachusetts General Hospital for two study visits over a 90-day window OR ability to access Zoom for virtual study visits
* Possess a smartphone
* Willingness to follow the study protocol

Exclusion Criteria:

* Presence of an MS relapse requiring acute management and/or hospitalization
* Daily medication provided by allied health care workers
* Foreign travel preventing electronic remote monitoring
* Expectation of discontinuation of the oral disease modifying therapy (DMT) in the upcoming 90 days for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
Rate of perfect adherence | 90-days post-enrollment
  Perfect adherence is defined as taking all scheduled pills +/-3 hours of scheduled dosing time

SECONDARY OUTCOMES:
Participant satisfaction | 90-days post-enrollment
  Participant satisfaction with the use of an electronic pill bottle and app

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Menzin J, Caon C, Nichols C, White LA, Friedman M, Pill MW. Narrative review of the literature on adherence to disease-modifying therapies among patients with multiple sclerosis. J Manag Care Pharm. 2013 Jan-Feb;19(1 Suppl A):S24-40. doi: 10.18553/jmcp.2013.19.s1.S24. PMID 23383731
- [Background] Schreiber K, Kant M, Pfleger C, Jensen HB, Oesterberg O, Hald AR, Nielsen FK, Rubak S. High treatment adherence, satisfaction, motivation, and health-related quality of life with fingolimod in patients with relapsing-remitting multiple sclerosis - results from a 24-month, multicenter, open-label Danish study. Patient Prefer Adherence. 2018 Jun 29;12:1139-1150. doi: 10.2147/PPA.S166278. eCollection 2018. PMID 29988735
- [Background] Erbay O, Usta Yesilbalkan O, Yuceyar N. Factors Affecting the Adherence to Disease-Modifying Therapy in Patients With Multiple Sclerosis. J Neurosci Nurs. 2018 Oct;50(5):291-297. doi: 10.1097/JNN.0000000000000395. PMID 30138155